CLINICAL TRIAL: NCT06562998
Title: Pentoxifylline Prophylactic Role Against Paclitaxel Chemotherapy-induced Neuropathy
Brief Title: Pentoxifylline Role Against Chemotherapy-induced Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Lecturer of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMBSUREC/07072024
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTX group (Active Comparator): paclitaxel based regimens plus Pentoxifylline 400mg twice daily for 12weeks.
  Interventions: Drug: Pentoxifylline
- Control group (Placebo Comparator): include those assigned for Taxol-based chemotherapy without intervention for 12 weeks
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400mg twice daily plus paclitaxel based regimens for 12weeks.

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and debilitating side effect of neurotoxic cancer treatment. Estimated to occur in up to 80% of paclitaxel-treated patients with breast cancer, neuropathy symptoms can interfere with function, increasing the risk of falls and reducing quality of life. To date, there are no approved medications for the prevention and/or treatment of CIPN. The objective of the present study is to investigate the beneficial effects of pentoxifylline (PTX) against CIPN in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients> 18 years old.
* Female patients Breast cancer patients who received paclitaxel-based regimen for 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance ≤ 2-Adequate bone marrow function.
* Adequate liver and kidney function.

Exclusion Criteria:

* Children less than 18 years old.
* Evidence of physical diseases or major surgery.
* Patientswith a history of chronic diseases including; renal, hepatic, gastrointestinal, respiratory, hematological, and metabolic or other diseases.
* Patients with preexisting clinical neuropathy.
* Patients with diabetes mellitus.
* Metastatic breast cancer.
* Patients receiving medications that ameliorate neuropathy like; antidepressants, anticonvulsants, opioids, adjuvant or topical analgesics.
* Patients treated with medications that increase the risk of neuropathy.
* Hypersensitivity to pentoxifylline or xanthine derivatives.
* Patients retinal bleeding or active peptic ulcer.
* Patients at high risk for bleeding or taking medications that increase risk of bleeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity(FACT-GOG-NTX) subscale | 12 weeks

SECONDARY OUTCOMES:
Common Terminology Criteria for Adverse Events Version 5 (CTCAE v5) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kidwani MA, Osama H, Hassan A, Abdelrahim MEA. Prophylactic role of pentoxifylline against paclitaxel-induced neuropathy among patients with breast cancer: a randomized-controlled trial. Anticancer Drugs. 2025 Feb 1;36(2):126-134. doi: 10.1097/CAD.0000000000001666. Epub 2024 Oct 16. PMID 39423312